CLINICAL TRIAL: NCT05919667
Title: The Effects of Dairy and Non-Dairy Alternatives on Glycemic and Appetite Regulation in Healthy Young Adults
Brief Title: Dairy and Non-Dairy Alternatives Comparative on Metabolic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MYC_AcuteDairy_2022
Record Dates: First submitted 2022-02-28; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: Dairy; Post-prandial glycemia; Appetite; Satiety; Gut Hormone Responses
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Polymethyl Methacrylate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomized, single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dairy-based Product 1 (Experimental): 2% Cow's milk (Neilson, St-Laurent, Quebec)
  Interventions: Dietary Supplement: Dairy and plant-based dairy beverages and solids
- Dairy-based Product 2 (Experimental): Regular fat cheddar cheese (Armstrong, St-Laurent, Québec)
  Interventions: Dietary Supplement: Dairy and plant-based dairy beverages and solids
- Plant-based Product 3: (Experimental): Vanilla Soy Beverage (Silk, Broomfield, Colorado)
  Interventions: Dietary Supplement: Dairy and plant-based dairy beverages and solids
- Plant-based Product 4 (Experimental): Vanilla Almond Beverage (Earth's Own, Vancouver, British Columbia)
  Interventions: Dietary Supplement: Dairy and plant-based dairy beverages and solids
- Plant-based Product 5 (Experimental): Plant-based Cheddar-Style Block (President' Choice, Brampton, Ontario)
  Interventions: Dietary Supplement: Dairy and plant-based dairy beverages and solids

INTERVENTIONS:
Dietary Supplement: Dairy and plant-based dairy beverages and solids — Crossover design: participants received all treatment arms in a randomized order

SUMMARY:
The purpose of this study is to compare the acute effects of a single serving of dairy and non-dairy alternatives on post-treatment and post-meal glycemia, appetite, plasma amino acid concentrations, and gastrointestinal hormones levels.

DETAILED DESCRIPTION:
In the past forty years, the prevalence of obesity in adults has doubled with nearly two thirds of Canadian adults currently overweight or obese. The global epidemic of obesity also makes certain individuals more vulnerable to common co-morbidities of obesity, such as type-2-diabetes. To combat these rising numbers, Health Canada released a new Canadian Food Guide (CFG) in 2019. One particular alteration to the new CFG includes dietary guidelines encouraging for an increased consumption of plant-based foods as protein rich sources, shifting away from the promotion of animal-based food products, such as dairy. However, many of the available plant-based substitutes in the market are highly processed with high amounts of sugar, fat, sodium, and additives compared to animal-based products. While literature has shown for plant-based foods to confer numerous health benefits, these are often plant-based foods that have been unprocessed, except for cooking. As the demand for plant-based products continues to grow annually, it is important to assess and compare various obesity and T2D related metabolic outcomes, such as glycemic regulation and appetite control, to better understand the physiological functionality of these products and what role they may or may not play in mitigating the obesity and T2D global epidemics. There is a growing body of evidence from clinical and meta-analysis trials that show dairy products reduce satiety and provide better glycemic control; highlighting their potential to help reduce risk factors associated with obesity and T2D. However, literature has mainly focused on nutrient profile or isolated protein comparatives between animal and plant-based sources. Instead, this study will be looking at comparing dairy products and their plant-based counterparts with respect to their food matrix as a whole, to understand what responses these products produce in the form consumers are naturally eating them by. This study will focus on assessing the metabolic outcomes related to satiety and glycemic regulation. Satiety is an important physiological function related to food intake, and thus, provides a measure to assess reduced obesity risk. Additionally, postprandial glycemic control is an important physiological function that is not only related to the development of type-2 diabetes but also satiety.

A total of 16 participants (8 males and 8 females) will participate in this study at the University of Toronto.

The study will include a total of 5 sessions over the span of 5 weeks. Prior to the visit, participants will be fasted for 12 hours, excluding water for up to 1 hour before the study visit. During each session, participants will consume a dairy product or a non-dairy plant-based product while subjective appetite, blood glucose, insulin, C-peptide, and gut hormones (ghrelin, GLP-1, GLP-2, and GIP) are obtained post-treatment at 20 min and post a secondary fixed meal of pasta within 15-30 min intervals over a 2 hour timespan. Plasma amino acid concentrations will also be measured within the same timeline outlined above.

ELIGIBILITY:
Inclusion Criteria:

* BMI: ≥18.5 kg/m2 and ≤ 24.5 kg/m2'
* Fasting serum glucose: ≤ 5.5 mmol/L
* Frequent breakfast consumers
* Willing to maintain habitual diet, physical activity pattern, dietary supplement routine, and body weight throughout the trial
* Willing to abstain from alcohol consumption for 24 h prior to all test visits.
* Willing to avoid vigorous physical activity for 24 h prior to all test visits.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Fasting blood glucose > 5.5 mmol/L
* Smoking tobacco products and marijuana regularly
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease
* Presence of gastrointestinal disorder or surgeries within the past year
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose, appetite and/or any other outcomes of the study as per investigator's judgment
* Known to be pregnant or lactating, or planning on becoming pregnant in the next 12 months
* Irregular menstrual cycles (i.e., frequent missed cycles), menopausal or post- menopausal
* Breakfast skippers
* Currently trying to lose or gain weight and any weight gain or loss of at least 10 lbs in previous three months
* Known intolerance, sensitivity or allergy to dairy products (including milk and cheese)
* Consumption of powders/protein supplements
* Extreme dietary habits
* Excessive alcohol intake
* Restrained Eaters

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose level | Starting at the beginning of each sessions (0 min, before consumption of treatment) and every 15-30 minutes up to 160 minutes]. A total of 9 times.
  Venous blood collection via catheter

SECONDARY OUTCOMES:
Subjective appetite | Measured every 15-30 minutes up to 160 minutes]. A total of 9 times.
  Quantifying appetite by using Visual Analogue Scales. Scored 0 to 100
  1. How strong is your desire to eat?
  2. How hungry do you feel?
  3. How full do you feel?
  4. How much food do you think you could eat?
Change in plasma metabolic and gut hormones (insulin, c-peptide, glucagon-like 1 receptor, glucagon-like 2 peptide and gastric inhibitory polypeptide) | Starting at the beginning of each session (0 minutes, before consumption of treatment) and every 15-30 minutes up to 160 minutes]. A total of 7 times.
  Venous blood collection via catheter
Change in plasma amino acid concentrations | Starting at the beginning of each session (0 minutes, before consumption of treatment) and every 15-30 minutes up to 160 minutes]. A total of 7 times.
  Venous blood collection via catheter

CONTACTS AND LOCATIONS:
Overall Officials: G. Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, C. David Naylor Building, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Da Silva N, Anderson G, Amr A, Vien S, Fabek H. A comparison of the effects of dairy products with their plant-based alternatives on metabolic responses in healthy young Canadian adults: a randomized crossover study. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-17. doi: 10.1139/apnm-2024-0158. PMID 39146559